CLINICAL TRIAL: NCT02606214
Title: A Phase I, Double-Blind, Placebo Controlled, Randomized, Multiple Ascending Dose Study With a Dose Formulation Comparison Cohort to Evaluate the Safety, Tolerability, and Pharmacokinetics of TBA-354 in Healthy Adult Subjects
Brief Title: A Multiple Ascending Dose Study With a Dose Formulation Comparison Cohort to Evaluate the Safety, Tolerability, and Pharmacokinetics of TBA-354 in Healthy Adult Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Clinical Hold from FDA
Sponsor: Global Alliance for TB Drug Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TBA-354-CL-002
Record Dates: First submitted 2015-11-05; First posted 2015-11-17 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; TBA-354; Pulmonary Tuberculosis; TB
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary | interventions — TBA-354

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Dose Level 1: 50 mg TBA-354 (Experimental): 50 mg TBA-354 for 14 days (two 25 mg once daily)
  Interventions: Drug: TBA-354
- Dose Level 1: Placebo (Placebo Comparator): Placebo cohort for Dose Level 1
  Interventions: Drug: TBA-354 Placebo
- Dose Level 2: 100 mg TBA-354 (Experimental): 100 mg TBA-354 for 14 days (one 100 mg tablet once daily)
  Interventions: Drug: TBA-354
- Dose Level 2: Placebo (Placebo Comparator): Placebo cohort for Dose Level 2
  Interventions: Drug: TBA-354 Placebo
- Dose Level 3: 200 mg TBA-354 (Experimental): 200 mg TBA-354 for 14 days (two 100 mg once daily)
  Interventions: Drug: TBA-354
- Dose Level 3: Placebo (Placebo Comparator): Placebo cohort for Dose Level 3
  Interventions: Drug: TBA-354 Placebo
- Dose Formulation Comparison Cohort (Experimental): All subjects in this cohort will receive two doses of the active drug. The first dose in three subjects will be a 100 mg TBA-354 tablet, followed 14 days later by a 100 mg dose of the TBA-354 suspension formulation. The first dose in the other three subjects will be 100 mgs of the TBA-354 suspension formulation, followed 14 days later by a 100 mg TBA-354 tablet dose. Placebo formulations will not be used in the dose formulation comparison cohort.
  Each dose will be administered orally with 200 ml of water after a minimum 8 hour overnight fast. Food will be given two hours after each dose.
  Interventions: Drug: TBA-354

INTERVENTIONS:
Drug: TBA-354
  Arms: Dose Formulation Comparison Cohort; Dose Level 1: 50 mg TBA-354; Dose Level 2: 100 mg TBA-354; Dose Level 3: 200 mg TBA-354
Drug: TBA-354 Placebo
  Arms: Dose Level 1: Placebo; Dose Level 2: Placebo; Dose Level 3: Placebo

SUMMARY:
The objective of the study is to evaluate the safety and tolerability of multiple doses of TBA-354 in healthy subjects.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multiple ascending dose study conducted at one study center in the United States. Three (3) multiple ascending dose cohorts are planned with twelve (12) healthy subjects (9 active and 3 placebo) in each cohort. There will also be a dose formulation comparison cohort, enrollment of six (6) subjects is planned. An additional multiple dose cohort of twelve (12) subjects may be enrolled.

Safety will be assessed throughout the study; serial ECGs and serial blood samples will be collected for the safety and pharmacokinetics (PK) assessment of TBA-354.

Dose escalation to the next cohort (i.e., dose level) will not take place until the Sponsor, in conjunction with the Principal Investigator, has determined that adequate safety, tolerability and PK from the previous cohort has been demonstrated to permit proceeding to the next cohort. Upon review of cohort data, the Sponsor, in conjunction with the Principal Investigator, may decide to:

1. Escalate the dose as planned.
2. Evaluate an intermediate dose level prior to proceeding to the next planned dose level if concerns arise from PK and safety that do not warrant in ceasing escalation.
3. Repeat a given dose level in a new cohort of subjects.
4. Increase the dose of the next cohort if the PK is lower than expected in the previous cohort.
5. Add a cohort if the PK is lower than expected after a cohort and there are no safety concerns.
6. Halt the study.

During dose escalation, at no time will the projected Cmax of any individual exceed 7.6 µg/mL, which is the highest mean value at the no-observed-adverse-effect-level from the 3-month log toxicology study TBA 354 NCLN-103. The predicted median Cmax of the final cohort can exceed 3.2 µg/mL only if there have been no safety concerns.

Subjects in the Multiple Ascending Dose (MAD) Cohorts will be housed in the Celerion clinic from check-in to Day 15. Subjects will return to the clinic each day from Day 16-Day 21 and have a final one-week follow up phone interview upon completion. Subjects in the Dose Formulation Cohort will be housed in the Clerion clinic from check-in to Day 3, visit the clinic each day for Days 4-7, and be housed in the clinic for Days 14-16. Then subjects will return for a daily visit for Days 17-20, and be contacted for a final one-week follow up phone interview upon completion on Day 28.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male and females of non-childbearing potential, 19 to 50 years of age (inclusive) at the time of screening.
2. Body mass index (BMI) ≥ 18.5 and ≤ 32.0 (kg/m2) and a body weight of no less than 50.0 kg.
3. Medically healthy with no clinically significant screening results (e.g., laboratory profiles, medical histories, vital signs, ECGs, physical examination) as deemed by the Investigator.
4. No use of tobacco or nicotine containing products (including smoking cessation products), for a minimum of 6 months prior to dosing.
5. Females of non-childbearing potential, having undergone one of the following sterilization procedures at least 6 months prior to dosing:

   * Hysteroscopic sterilization
   * Bilateral tubal ligation or bilateral salpingectomy
   * Hysterectomy
   * Bilateral oophorectomy
   * or be postmenopausal with amenorrhea for at least 1 year prior to the first dose with serum follicle stimulating hormone (FSH) levels consistent with postmenopausal status at screening.
6. Non-vasectomized males (or males vasectomized less than 120 days prior to study start), must agree to the following during study participation and for 90 days following the last administration of study drug:

   * use a condom with spermicide while engaging in sexual activity or be sexually abstinent
   * not donate sperm during this time.

   In the event the sexual partner is surgically sterile, use of a condom with spermicide is not necessary. None of the restrictions listed above are required for vasectomized males whose procedure was performed more than 120 days prior to study start.
7. Willing to answer inclusion and exclusion criteria questionnaire at check-in.
8. Subject understands study procedures and provides written informed consent for the trial.
9. Be able to comply with the protocol and the assessments therein, including all restrictions.

Exclusion Criteria:

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease as determined by the Investigator to be clinically relevant.
2. History of any illness that, in the opinion of the Investigator, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
3. Surgery within the past 90 days prior to dosing as determined by the Investigator to be clinically relevant.
4. History or presence of alcoholism or drug abuse within the past 2 years as determined by the Investigator to be clinically relevant.
5. Hypersensitive or idiosyncratic reactions to compounds related to TBA-354 (e.g., nitroimidazoles such as metronidazole, etc.).
6. Female subjects who are pregnant or lactating.
7. Positive results for the urine drug/alcohol screen at screening or check-in.
8. Positive urine cotinine at screening.
9. Serum magnesium potassium, or calcium laboratory values outside of the normal range at screening.
10. Positive results at screening for Human Immunodeficiency Virus (HIV), Hepatitis B Surface Antigen (HBsAg), or Hepatitis C antibodies (HCV).
11. Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at screening.
12. Heart rate is lower than 40 bpm or higher than 99 bpm at screening.
13. Any electrocardiogram abnormality at Screening (as deemed by decision of the Investigator and the Sponsor's Medical Monitor).

    NOTE: The following can be considered not clinically significant without consulting the Sponsor's Medical Monitor:
    * Mild first degree A-V block (P-R interval <0.23 sec)
    * Right or left axis deviation
    * Incomplete right bundle branch block
    * Isolated left anterior fascicular block (left anterior hemiblock) in younger athletic subjects
14. QTcF interval >450 msec for males or >470 msec for females at screening, Day -2, Day -1, or Day 1 (pre-dose), or history of prolonged QT syndrome.
15. Family history of Long-QT Syndrome or sudden death without a preceding diagnosis of a condition that could be causative of sudden death (such as known coronary artery disease, congestive heart failure or terminal cancer).
16. History of one or any combination of, the following:

    * Seizures or seizure disorders
    * Brain surgery.
    * History of head injury in the last five years
    * Any serious disorder of the CNS or related neurological system, particularly one that may lower the seizure threshold. v. History of seizures
17. Use of any prescription medication within 14 days prior to dosing.
18. Use of any over-the-counter (OTC) medication, including herbal products and vitamins, within the 7 days prior to dosing, except acetaminophen. Up to 3 grams per day of acetaminophen is allowed at the discretion of the Investigator prior to dosing.
19. Use of any drugs or substances known to be significant inhibitors of Cytochrome P450 (CYP) enzymes and/or significant inhibitors or substrates of P-glycoprotein (P-gp) and/or Organic anion transporting polypeptides (OATP) within 14 days prior to the first dose of study drug.
20. Use of any drugs or substances known to be inducers of CYP enzymes and/or P-gp, including St. John's Wort, within 28 days prior to the first dose of study drug.
21. Use of any drugs or substance known to lower the seizure threshold.
22. Blood donation or significant blood loss within 56 days prior to dosing.
23. Plasma donation within 7 days prior to dosing.
24. Participation in another clinical trial within 28 days prior to dosing.
25. Prior treatment with investigational products pretomanid or OPC-67683.
26. Consumption of the following prior to dosing period:

    * Alcohol 48 hours prior to dosing
    * Grapefruit/Oranges 10 days prior to dosing
    * Caffeine/Xanthine 24 hours prior to dosing

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-11; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The comparison of the percentage of subjects per dose cohort with treatment emergent adverse events (TEAEs) from Days 1 to 28 compared to placebo | Multiple Ascending Dose Cohorts: Days 1-28, Dose Formulation Cohort: Days 1-28
The percent of subjects per cohort with safety electrocardiogram change-from-baseline QTcF intervals of >30 milliseconds and =>60 milliseconds. | Multiple Ascending Dose Data Time Point Days 1-3, 8, 12, 14-15, 21; Dose Formulation Cohort Data Time Point Days 1-3,7,14-16, 20
  QTcF = QT interval correct by Fridericia's method, percent = number of events/number of subjects

SECONDARY OUTCOMES:
The mean Tmax of TBA-354 per dose cohort in plasma following dosing | Multiple Ascending Dose Cohort: Days 1-14, Dose Formulation Cohort: Days 1-20
  Acronyms: Tmax = Time of the maximum drug concentration (obtained without interpolation).
The mean Cmax of TBA-354 per dose cohort in plasma following dosing | Multiple Ascending Dose Cohort: Days 1-14, Dose Formulation Cohort: Days 1-20
  Acronyms: Cmax= Maximum observed drug concentration
The mean AUC0-24 of TBA-354 per dose cohort in plasma following dosing | Multiple Ascending Dose Cohort: Days 1-14, Dose Formulation Cohort: Days 1-20
  Acronyms: AUC0-24= Area under concentration time curve 0 to 24 hours